CLINICAL TRIAL: NCT04954352
Title: Epidemiology in Humans of New Arbovirusus Sorted Out From Metagenomic Screen in Local Vectors and Animal Hosts.
Brief Title: Human Epidemiology of Newly Identified Arboviruses
Acronym: ARBODOCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: UMR ASTRE (CIRAD) (Unknown); Institut Pasteur (Industry); UMR PCCEI (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0297
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Arbovirus Infections; SARS-CoV Infection
Keywords: Patients with arboviral infection compatible signs; Unexplained isolated fever; Neurological infection conditions without any identified etiology; Arbovirus; Arboviral like infectious disease
MeSH Terms: conditions — Arbovirus Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood and CSF samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A local network is being set up to study the impact of arboviruses in our region. It is committed to a one-health approach, in particular with research without a priori for new viruses hosted among vectors and wildlife. The candidates identified by high throughput sequencing approaches will serve as a basis for the development of serological and molecular tools for their detections. These tools will be used to assess the possible circulation of these new viruses in humans in biological collections created within the framework of this project Arbodocc

.

ELIGIBILITY:
Inclusion criteria:

- Patients admitted at the Monpellier University Hospital for any infectious syndrome compatible with an arboviral infection with samples available

Exclusion criteria:

- Informed consent non obtain for samples used

Max Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * Patients admitted at the Monpellier University Hospital for any infectious syndrome compatible with an arboviral infection
  * Healthy volunteers for seroprevalence investigation
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Seroprevalence | 1 day
  Detection of antibodies targeting specific antigens of newly identified arboviruses

SECONDARY OUTCOMES:
Molecular detection | 1 day
  Detection of newly identified arboviruses genome

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Foulongne, PhD, Study Director — UH MONTPELLIER
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC